CLINICAL TRIAL: NCT00499525
Title: A Double-Blind, Randomized Phase 2b Study Evaluating the Efficacy and Safety of Sorafenib Compared to Placebo When Administered in Combination With Paclitaxel in Patients With Locally Recurrent or Metastatic Breast Cancer
Brief Title: Phase 2b Study of Taxol Plus Sorafenib or Placebo in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NU 07B1; NU 07B1 (Other: Northwestern University); STU00000776 (Other: Northwestern University IRB)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Paclitaxel; Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive paclitaxel IV over 1 hour once weekly for 3 weeks. Patients also receive oral sorafenib tosylate twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Drug: sorafenib tosylate
- Arm II (Active Comparator): Patients receive paclitaxel as in arm I and oral placebo twice daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: paclitaxel; Other: placebo

INTERVENTIONS:
Drug: paclitaxel — given IV
Drug: sorafenib tosylate — given orallly
  Arms: Arm I
Other: placebo — given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving paclitaxel together with sorafenib may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well paclitaxel works when given together with or without sorafenib in treating patients with locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare progression-free survival of patients with locally recurrent or metastatic breast cancer treated with sorafenib tosylate and paclitaxel versus placebo and paclitaxel as first-line therapy.

Secondary

* Compare the objective response rate and duration of response in patients treated with these regimens.
* Compare the time to progression in patients treated with these regimens.
* Compare the survival of patients treated with these regimens.
* Compare the safety of patients treated with these regimens.
* Compare the change from baseline in the Functional Assessment of Cancer Therapy for Breast Cancer quality of life assessment score in patients treated with these regimens.

OUTLINE: This is a double-blind, randomized, multicenter study. Patients are stratified according to site of metastatic disease (visceral [i.e., soft internal organs of the body, including lungs, heart, and the organs of the digestive, excretory, and reproductive systems] vs nonvisceral [i.e., osseous or soft tissue] sites). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive paclitaxel IV over 1 hour once weekly for 3 weeks. Patients also receive oral sorafenib tosylate twice daily on days 1-28.
* Arm II: Patients receive paclitaxel as in arm I and oral placebo twice daily on days 1-28.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, and every 8 weeks for 24 weeks, and then every 12 weeks for the duration of study participation.

After completion of study therapy, patients are followed every 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Locally recurrent or metastatic disease

    * Locally recurrent disease not amenable to resection with curative intent
* Measurable or evaluable disease
* No HER-2 overexpression (defined as positive for gene amplification by FISH or 3+ overexpression by IHC)

  * No unknown HER-2 status
* No active brain metastases

  * Patients with neurological symptoms and known brain metastases treated with definitive therapy must undergo contrast CT scan or brain MRI to exclude active brain metastasis

    * Previously treated brain metastases allowed provided at least 3 months since prior definitive therapy (including steroids) AND no evidence of disease
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* ECOG performance status 0-1
* Not pregnant or nursing for ≥ 2 weeks after completion of study therapy
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 2 weeks after completion of study therapy
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
* ALT and AST ≤ 2.5 times ULN (≤ 5 times ULN for patients with liver involvement)
* INR ≤ 1.5 and aPTT within normal limits

  * Anticoagulation therapy (e.g., warfarin or heparin) allowed

    * Stable INR required for patients on warfarin
* Creatinine ≤ 1.5 times the ULN
* Able to swallow and retain oral medication
* More than 4 weeks since prior significant traumatic injury
* No evidence or history of bleeding diathesis or coagulopathy
* No serious nonhealing wound, ulcer, or bone fracture
* No substance abuse or medical, psychological, or social condition that would interfere with study participation or evaluation of study results
* No pre-existing peripheral neuropathy ≥ grade 2
* No clinically significant cardiac disease, including any of the following:

  * New York Heart Association class II-IV congestive heart failure
  * Unstable angina (i.e., angina symptoms at rest) or new-onset angina within the past 3 months
  * Myocardial infarction within the past 6 months
* No cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 90 mm Hg despite optimal medical management)
* No thrombolic, embolic, venous, or arterial events such as a cerebrovascular accident, including transient ischemic attacks within the past 6 months
* No pulmonary hemorrhage or bleeding event > grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ grade 3 within the past 4 weeks
* No active clinically serious infection > grade 2
* No known HIV infection or chronic hepatitis B or C
* No other prior or concurrent cancer except carcinoma in situ of the cervix, treated basal cell skin cancer, superficial bladder tumors (e.g., Ta and Tis), or any cancer curatively treated for > 5 years
* No known or suspected allergy to sorafenib tosylate or hypersensitivity to paclitaxel or drugs using the vehicle Cremophor

PRIOR CONCURRENT THERAPY:

* More than 12 months since prior adjuvant or neoadjuvant taxane therapy
* At least 3 weeks since other prior adjuvant chemotherapy
* At least 3 weeks since prior hormonal therapy for locally recurrent or metastatic disease
* No prior chemotherapy for locally recurrent or metastatic breast cancer
* More than 4 weeks since prior major surgery or open biopsy
* At least 3 weeks since prior radiotherapy

  * Previously irradiated area must not be the only site of disease
* More than 30 days or 5 half-lives, whichever is longer, since prior investigational drug

  * No prior or concurrent bevacizumab or any other licensed or investigational drugs that target VEGF or VEGF-receptor
* More than 3 weeks since prior and no concurrent Hypericum perforatum (St. John's wort ) or rifampin (rifampicin)
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent irinotecan hydrochloride or doxorubicin hydrochloride
* No other concurrent anticancer therapy (i.e., chemotherapy, radiotherapy, surgery, immunotherapy, biologic therapy, or tumor embolization)
* No concurrent nonconventional therapies (e.g., herbal)
* No concurrent palliative radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-06; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | At disease progression or death

SECONDARY OUTCOMES:
Overall survival | At time of death
Time to progression | At time of disease progression
Overall response rate | At the time of progression of disease
Duration of overall response | At time of disease progression
Treatment-emergent adverse events as assessed by NCI CTCAE v3.0 | During treatment and up to 30 days post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (43):
- United States (43):
  - Northwest Alabama Cancer Center, PC - Muscle Shoals, Muscle Shoals, Alabama
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Pacific Cancer Medical Center, Incorporated, Anaheim, California
  - Pacific Coast Hematology/Oncology Medical Group, Incorporated, Fountain Valley, California
  - Desert Hematology-Oncology Medical Group, Incorporated, Rancho Mirage, California
  - Sutter Cancer Center, Sacramento, California
  - Cancer Prevention and Treatment Center at Dominican and Watsonville Community Hospital, Soquel, California
  - St. Helena, California
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Medical Oncology and Hematology, PC at Harold Leever Cancer Center, Waterbury, Connecticut
  - George Washington University Cancer Institute, Washington D.C., District of Columbia
  - Pasco Hernando Oncology Associates, PA - Brooksville, Brooksville, Florida
  - Pasco Hernando Oncology Associates, PA - New Port Richey, New Port Richey, Florida
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Hematology-Oncology Associates of Illinois, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cancer Institute at Alexian Brothers, Elk Grove Village, Illinois
  - Medical and Surgical Specialists, LLC, Galesburg, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Kellogg Cancer Care Center, Oak Park, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Family Medicine of Vincennes Clinical Trial Center, Vincennes, Indiana
  - Kentuckiana Cancer Institute, PLLC, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, Columbia, Missouri
  - Nebraska Hematology-Oncology, PC, Lincoln, Nebraska
  - Essex Oncology of North Jersey, Belleville, New Jersey
  - Sussex County Medical Associates - Sparta, Sparta, New Jersey
  - Piedmont Hematology-Oncology Associates, Winston-Salem, North Carolina
  - Tri-County Hematology/Oncology Associates, Incorporated, Canton, Ohio
  - Hematology Oncology Consultants, Incorporated, Columbus, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Hematology and Oncology Associates of Rhode Island, Cranston, Rhode Island
  - West Clinic - East Memphis, Memphis, Tennessee
  - Patients' Comprehensive Cancer Center - Carrollton, Carrollton, Texas
  - Oncology Consultants - Memorial City, Houston, Texas
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin